CLINICAL TRIAL: NCT00388505
Title: A Randomized, Open-label Multicentre Phase 3 Trial to Assess the Safety of Tobramycin Inhalation Powder Compared to Tobramycin Solution for Inhalation in Cystic Fibrosis Subjects
Brief Title: Safety of Tobramycin Inhalation Powder (TIP) vs Tobramycin Solution for Inhalation in Patients With Cystic Fibrosis
Acronym: EAGER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTBM100C2302
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Results first posted 2012-07-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-06

CONDITIONS: Cystic Fibrosis
Keywords: tobramycin
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation

ARMS (2):
- Tobramycin inhalation powder (TIP) (Experimental): Participants received four 28 mg capsules of tobramycin inhalation powder (TIP) delivered with the T-326 inhaler twice daily for 28 days followed by 28 days off therapy (one cycle) for a total of three cycles.
  Interventions: Drug: Tobramycin Inhalation Powder
- Tobramycin solution for inhalation (TOBI) (Active Comparator): Participants received one 300 mg (in 5 mL) ampoule of tobramycin solution for inhalation (TOBI) delivered with a nebulizer twice daily for 28 days followed by 28 days off therapy (one cycle) for a total of three cycles.
  Interventions: Drug: Tobramycin Solution for Inhalation

INTERVENTIONS:
Drug: Tobramycin Inhalation Powder — Tobramycin Inhalation Powder (TIP) capsules for inhalation.
  Arms: Tobramycin inhalation powder (TIP)
Drug: Tobramycin Solution for Inhalation — Tobramycin solution for inhalation (TOBI), supplied as 300 mg/5mL ampoules administered with a nebulizer
  Arms: Tobramycin solution for inhalation (TOBI)

SUMMARY:
This study compares the safety of the tobramycin solution for inhalation with the tobramycin dry powder formulation, used with a simple inhaler

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cystic fibrosis
* Male and female patients at least 6 years of age at the time of screening.
* Forced expiratory volume in one second (FEV1) at screening must be at least 25% and less than or equal to 75% of normal predicted values for age, sex, and height based on Knudson criteria.
* Pseudomonas aeruginosa, a type of bacteria, must be present in a sputum/deep-throat cough swab culture (or bronchoalveolar lavage [BAL]) within 6 months prior to screening and in the sputum/ deep-throat cough swab culture at the screening visit.
* Able to comply with all protocol requirements.
* Clinically stable in the opinion of the investigator.
* Use of an effective means of contraception in females of childbearing potential.
* Provide written informed consent, Health Authority Portability and Accountability Act (HIPAA) authorization (where applicable), and assent (as appropriate) prior to the performance of any study-related procedure.

Exclusion Criteria:

* History of sputum culture or deep-throat cough swab (or BAL) culture yielding Burkholderia cepacia (B cepacia), a type of bacteria, within 2 years prior to screening and/or sputum culture yielding B cepacia at screening.
* Coughing up more than 60 cc of blood from the respiratory tract at any time within 30 days prior to study drug administration.
* Known local or systemic hypersensitivity to aminoglycosides or inhaled antibiotics.
* Females who are pregnant (positive pregnancy test), lactating, or are planning to become pregnant during the study.
* History of hearing loss or chronic ringing in the ears deemed clinically significant by the investigator.
* Use of systemic or inhaled antipseudomonal antibiotics within 28 days prior to study drug administration.
* Use of loop diuretics within 7 days prior to study drug administration.
* Use of any investigational treatment within 28 days prior to study drug administration.
* Initiation of treatment with chronic macrolide therapy, dornase alpha treatment or inhaled corticosteroids within 28 days prior to study drug administration (patients may be taking these therapies at the time of enrollment, but they must have initiated treatment more than 28 days prior to study drug administration).

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Konstan, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (72):
- United States (24):
  - Novartis Investigative Site, Hartford, Connecticut
  - Emory University CF Center, Atlanta, Georgia
  - Rush University Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Livingston, New Jersey
  - Novartis Investigative Site, Long Branch, New Jersey
  - Novartis Investigative Site, Morristown, New Jersey
  - Novartis Investigative Site, Somerset, New Jersey
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New Hyde Park, New York
  - Novartis Investigative Site, New York, New York
  - University of Rochester, Rochester, New York
  - Novartis Investigative Site, Stony Brook, New York
  - Novartis Investigative Site, Syracuse, New York
  - Novartis Investigative Site, Valhalla, New York
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - West Virginia University Health Sciences Center, Morgantown, West Virginia
- Novartis Investigative Site, South Brisbane, Australia
- Canada (4):
  - Novartis Investigative Site, Calgary
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Ste-Foy
  - Novartis Investigative Site, Vancouver
- Novartis Investigative Site, Santiago, Chile
- Colombia (4):
  - Novartis Investigative Site, Baranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
  - Novartis Investigative Site, Medellín
- France (3):
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
- Germany (11):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Klinikum der Johann-Wolfgang-Goethe-Universitaet, Frankfurt
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Ludwig-Maximilians-Universitaet, Munich
  - Novartis Investigative Site, München
- Hungary (2):
  - Novartis Investigative Site, Hungary
  - Novartis Investigative Site, Kaposvár
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
- Italy (4):
  - Novartis Investigator Site, Genoa
  - Novartis Investigative Site, Palermo
  - Novartis Investigative Site, Potenza
  - Novartis Investigative Site, Roma
- Novartis Investigative Site, Monterrey Nuevo Leon, Mexico
- Netherlands (2):
  - Novartis Investigative Site, Groesbeek
  - Novartis Investigative Site, Rotterdam
- Spain (6):
  - Novartis Investigative Site, Barakaldo
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- United Kingdom (6):
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Sheffield

REFERENCES:
- See also: Related Info — http://www.novartisclinicaltrials.com/webapp/etrials/home.do

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Started | 308 (Randomized patients who received any amount of study medication) | 209 (Randomized patients who received any amount of study medication)
Completed | 225 | 171
Not Completed | 83 | 38
Not completed — Adverse Event or Death | 43 | 17
Not completed — Withdrawal by Subject | 24 | 9
Not completed — Lost to Follow-up | 5 | 3
Not completed — Inappropriate Enrollment | 0 | 1
Not completed — Administrative Reason | 1 | 0
Not completed — Protocol Violation | 6 | 5
Not completed — Unable to classify | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI) | Total
Number analyzed (Participants) | 308 | 209 | 517
Age Continuous [Mean (Standard Deviation); unit: years] | 25.9 (11.36) | 25.2 (10.20) | 25.6 (10.90)
Age, Customized [Number; unit: participants]
  ≥6 to <13 years | 28 | 18 | 46
  ≥13 to <20 years | 66 | 48 | 114
  ≥20 years | 214 | 143 | 357
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 94 | 231
  Male | 171 | 115 | 286

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence, including any unfavorable and unintended sign, symptom or disease temporally associated with the use of the study medication that does not necessarily have a causal relationship with study medication. A serious AE (SAE) is an event that results in death, is life-threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability, is a congenital anomaly or defect, or is a significant medical event that may jeopardize the patient or require intervention to prevent one of the outcomes listed above.
Time Frame: 25 weeks
Population: All Randomized Safety population.
Measure: Number; unit: participants
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Number analyzed (Participants) | 308 | 209
participants
  Any adverse event | 278 | 176
  Serious adverse event | 85 | 61
  Death | 3 | 0
  Discontinued due to AE(s) | 46 | 17
  Discontinued due to SAE(s) | 14 | 6

2. Secondary Outcome: Serum Tobramycin Concentrations
Description: Serum tobramycin concentrations were measured in a subset of participants at Week 1 (start of cycle 1), Week 5 (End of Cycle 1), Week 17 (start of cycle 3) and Week 21 (end of cycle 3). Serum samples were collected at pre-dose and post-dose at specified intervals; one specimen between 0 to 2 hours; two additional specimens between 2 and 5 hours (sample times must have been a minimum of 2 hours apart).
Time Frame: Weeks 1, 5, 17 and 21
Population: Pharmacokinetic subpopulation
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Number analyzed (Participants) | 28 | 14
μg/mL
  Week 1: Predose [N=28, 14] | 0.00 (0.02) | 0.02 (0.05)
  Week 1: 0 to 2 hours [N=28, 14] | 0.82 (0.39) | 0.61 (0.35)
  Week 1: 2 to 5 hours (1st sample) [N=26, 14] | 0.74 (0.34) | 0.69 (0.39)
  Week 1: 2 to 5 hours (2nd sample) [N=25, 12] | 0.68 (0.24) | 0.54 (0.25)
  Week 5: Predose [N=23, 13] | 0.47 (0.73) | 0.21 (0.15)
  Week 5: 0 to 2 hours [N=23, 12] | 1.39 (0.80) | 1.18 (0.72)
  Week 5: 2 to 5 hours (1st sample) [N=23, 11] | 1.41 (0.60) | 1.08 (0.55)
  Week 5: 2 to 5 hours (2nd sample) [N=23, 8] | 1.09 (0.50) | 0.83 (0.34)
  Week 17: Predose [N=24, 13] | 0.07 (0.22) | 0.08 (0.25)
  Week 17: 0 to 2 hours [N=24, 13] | 0.75 (0.54) | 0.87 (0.54)
  Week 17: 2 to 5 hours (1st sample) [N=24, 12] | 0.80 (0.34) | 0.91 (0.64)
  Week 17: 2 to 5 hours (2nd sample) [N=23, 12] | 0.74 (0.30) | 0.67 (0.40)
  Week 21: Predose [N=24, 13] | 0.36 (0.29) | 0.24 (0.26)
  Week 21: 0 to 2 hours [N=24, 12] | 1.22 (0.57) | 1.10 (0.64)
  Week 21: 2 to 5 hours (1st sample) [N=22, 12] | 1.19 (0.50) | 1.02 (0.52)
  Week 21: 2 to 5 hours (2nd sample) [N=24, 11] | 1.03 (0.36) | 0.84 (0.40)

3. Secondary Outcome: Percentage of Participants With a Decrease From Baseline in Auditory Acuity
Description: Audiology testing was performed only at selected centers. Auditory acuity was measured from 250 to 8000 Hertz using a standard dual-channel audiometer.
Time Frame: Baseline and Day 28 of Cycles 1, 2 and 3 (Weeks 5, 13 and 21)
Population: Audiology subpopulation
Measure: Number; unit: percentage of participants
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Number analyzed (Participants) | 73 | 42
percentage of participants
  Cycle 1, Day 28 [N=60, 39] | 13.3 | 10.3
  Cycle 2, Day 28 [N=55, 34] | 12.7 | 0.0
  Cycle 3, Day 28 [N=54, 34] | 18.5 | 11.8

4. Secondary Outcome: Relative Change From Baseline in Percent Predicted Forced Expiratory Volume in One Second (%FEV1)
Description: Forced expiratory volume in one second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 is then converted to a percentage of normal (percent predicted) based on height, weight, and race. FEV1 was measured at Baseline (prior to beginning study treatment) and predose on Day 28 of Cycles 1, 2 and 3 and at the follow-up visit.
  Relative change = 100 * ((Day 28 of Cycle 3 value - Baseline value)/ Baseline value).
Time Frame: Baseline and Day 28 of Cycles 1, 2 and 3 (Weeks 5, 13 and 21) and Final Visit (Week 25)
Population: Intent to treat population for patients with available data. For Final Visit, the last available post-baseline measurement is reported.
Measure: Mean (Standard Deviation); unit: percent of predicted
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Number analyzed (Participants) | 308 | 209
percent of predicted
  Baseline [N=308, 209] | 52.9 (14.20) | 52.8 (15.95)
  Change from Baseline at Week 5 [N=268, 194] | 2.8 (19.64) | 3.6 (14.33)
  Change from Baseline at Week 13 [N=252, 178] | 2.3 (18.76) | 4.3 (16.63)
  Change from Baseline at Week 21 [N=227, 171] | 3.1 (19.92) | 2.3 (17.57)
  Change from Baseline: Final Visit [N=307, 209] | -0.4 (17.15) | -1.6 (17.38)

5. Secondary Outcome: Patient Satisfaction Assessed Using the Treatment Satisfaction Questionnaire for Medication
Description: Patient's self-reported treatment satisfaction was measured using the Treatment Satisfaction Questionnaire for Medication (TSQM, a validated instrument) which was modified by adding four study-specific questions; the standard fourteen questions of the TSQM were not altered. Responses to nearly all items are rated on a five-point or seven-point rating scale and the items are factored into 4 domains. The TSQM domain scores range from 0 to 100 with higher scores representing higher satisfaction for that domain.
Time Frame: Day 28 of Cycles 1, 2 and 3 (Weeks 5, 13 and 21).
Population: Intent-to-treat population for whom data were available.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Number analyzed (Participants) | 308 | 209
Scores on a scale
  Cycle 1: Effectiveness [N=264, 189] | 74.1 (17.29) | 64.6 (18.63)
  Cycle 1: Side Effects [N=263, 190] | 92.1 (15.58) | 92.4 (15.99)
  Cycle 1: Convenience [N=264, 190] | 82.3 (14.95) | 58.1 (20.64)
  Cycle 1: Global Satisfaction [N=264, 190] | 75.4 (20.19) | 20.19 (18.67)
  Cycle 2: Effectiveness [N=241, 170] | 74.5 (17.62) | 64.6 (17.42)
  Cycle 2: Side Effects [N=239, 170] | 93.6 (14.06) | 93.8 (13.41)
  Cycle 2:Convenience [N=241, 170] | 81.1 (16.61) | 57.0 (20.40)
  Cycle 2: Global Satisfaction [N=241, 170] | 76.6 (19.16) | 70.2 (19.40)
  Cycle 3: Effectiveness [N=221, 162] | 74.9 (20.25) | 65.5 (17.42)
  Cycle 3: Side Effects [N=215, 158] | 91.5 (17.78) | 94.1 (14.48)
  Cycle 3: Convenience [N=221, 162] | 81.6 (16.89) | 56.6 (20.90)
  Cycle 3: Global Satisfaction [N=221, 162] | 75.2 (24.00) | 72.2 (17.90)

6. Secondary Outcome: Change From Baseline in Pseudomonas Aeruginosa Sputum Density
Description: Three Pseudomonas aeruginosa biotypes were assessed in patient's sputum; mucoid, dry and small colony variant. Overall density is defined as the sum of all bio-types in Pseudomonas aeruginosa density.
Time Frame: Baseline and Day 28 of Cycles 1, 2 and 3 (Weeks 5, 13 and 21) and Final Visit (Week 25).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 Colony forming units/g
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Number analyzed (Participants) | 308 | 209
log10 Colony forming units/g
  Baseline [N=279, 192] | 7.23 (1.49) | 7.35 (1.54)
  Change from Baseline at Week 5 [N=202, 145] | -1.76 (1.96) | -1.32 (2.03)
  Change from Baseline at Week 13 [N=170, 125] | -1.54 (1.99) | -1.11 (1.91)
  Change from Baseline at Week 21 [N= 157, 126] | -1.61 (2.03) | -0.77 (1.78)
  Change from Baseline: Final Visit [N=263, 179] | -0.53 (1.92) | -0.33 (1.71)

7. Secondary Outcome: Change From Baseline in Tobramycin Minimum Inhibitory Concentration
Description: The minimum inhibitory concentration (MIC) is the lowest concentration of an antimicrobial that will inhibit the visible growth of a microorganism after overnight incubation. The MIC of tobramycin against total Pseudomonas aeruginosa colonization was assessed over the course of the study.
Time Frame: Baseline and Day 28 of Cycles 1, 2 and 3 (Weeks 5, 13 and 21) and Final Visit (Week 25)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Number analyzed (Participants) | 308 | 209
μg/mL
  Baseline [N=308, 208] | 35.39 (107.58) | 42.45 (116.40)
  Change from Baseline at Week 5 [N=239, 173] | 38.47 (148.34) | 5.80 (112.96)
  Change from Baseline at Week 8 [N=215, 157] | 35.59 (148.03) | 20.68 (130.57)
  Change from Baseline at Week 21 [N=199, 154] | 29.83 (139.85) | 14.13 (117.54)
  Change from Baseline: Final Visit [N=298, 202] | 30.89 (139.63) | 3.27 (107.80)

8. Secondary Outcome: Antipseudomonal Antibiotic Usage During the Study
Description: The average number of days patients required antipseudomonal antibiotics during the course of the study.
Time Frame: 25 Weeks
Population: Patients in the intent-to-treat population who required antipseudomonal antibiotics.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Number analyzed (Participants) | 202 | 115
days | 34.5 (31.24) | 40.1 (37.27)

9. Secondary Outcome: Hospitalization Due to Respiratory Events During the Study
Description: The average number of days patients were hospitalized due to respiratory events during the course of the study.
Time Frame: 25 Weeks
Population: Patients in the intent-to-treat population who were hospitalized due to respiratory events.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Number analyzed (Participants) | 75 | 46
days | 15.6 (13.31) | 15.3 (10.23)

ADVERSE EVENTS:
Arm/Group | Tobramycin Inhalation Powder (TIP) | Tobramycin Solution for Inhalation (TOBI)
Serious Adverse Events (participants affected / at risk) | 85/308 | 61/209
Other Adverse Events (participants affected / at risk) | 241/308 | 148/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Powder (TIP) (N=308) | Tobramycin Solution for Inhalation (TOBI) (N=209)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Distal ileal obstruction syndrome (Gastrointestinal disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatic insufficiency (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Pyrexia (General disorders) | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 6 | 1
Bronchopneumonia (Infections and infestations) | 1 | 2
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Lung abscess (Infections and infestations) | 1 | 1
Lung infection pseudomonal (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 2
Pneumonia bacterial (Infections and infestations) | 2 | 2
Pseudomonas bronchitis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 1
Forced expiratory volume decreased (Investigations) | 1 | 1
Oxygen saturation (Investigations) | 1 | 0
Pulmonary function test decreased (Investigations) | 4 | 3
Weight decreased (Investigations) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 60 | 39
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Powder (TIP) (N=308) | Tobramycin Solution for Inhalation (TOBI) (N=209)
Abdominal pain (Gastrointestinal disorders) | 12 | 17
Nausea (Gastrointestinal disorders) | 23 | 19
Vomiting (Gastrointestinal disorders) | 19 | 11
Chest discomfort (General disorders) | 20 | 6
Fatigue (General disorders) | 18 | 10
Pyrexia (General disorders) | 47 | 25
Sinusitis (Infections and infestations) | 17 | 15
Upper respiratory tract infection (Infections and infestations) | 21 | 18
Pulmonary function test decreased (Investigations) | 18 | 14
Headache (Nervous system disorders) | 34 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 145 | 63
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 42 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 22
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 35 | 23
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 57 | 33
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 25 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 43 | 22
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 17 | 8
Rales (Respiratory, thoracic and mediastinal disorders) | 21 | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 22 | 15
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 49 | 35
Wheezing (Respiratory, thoracic and mediastinal disorders) | 21 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.